CLINICAL TRIAL: NCT03783169
Title: SASH Study - Sonographic Assessment for Severe Hypertension in Pregnancy
Acronym: SASH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 18-027
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic patients: All pregnant women (under the care of the Maternal-Fetal Medicine physicians or Faculty Medical Center physicians with MFM involvement) experiencing a hypertensive emergency (sustained systolic blood pressure > 160 mmHg or sustained diastolic blood pressure > 110 mmHg {or both} on at least two consecutive occasions 15 minutes apart). All participants must be over the age of 18 and capable of consenting to the study (conscious, with capacity for medical decision making for themselves).
  Interventions: Other: Cardiovascular Sonographic Assessment
- Asymptomatic patients: All asymptomatic pregnant women who are undergoing routine obstetric ultrasound evaluations at any gestational age who elect to undergo cardiovascular sonographic assessment for research purposes at no cost. All participants must be over the age of 18 and capable of consenting to the study (conscious, with capacity for medical decision making for themselves).
  Interventions: Other: Cardiovascular Sonographic Assessment

INTERVENTIONS:
Other: Cardiovascular Sonographic Assessment — Maternal sonographic vascular measurements assessing volume status, cardiac output, and systemic vascular resistance by means of inferior vena cava collapsibility/caval index (ICV CI), end-point septal separation (EPSS) for determining left ventricular ejection fraction (LVEF), cardiac output determination (stroke volume x heart rate), stroke volume variation, & radial artery resistance index) augments standard vital sign assessment (pulse pressure and systolic / diastolic predominance)

SUMMARY:
• Adjunctive use of easily-obtainable maternal sonographic vascular measurements assessing volume status, cardiac output, and systemic vascular resistance by means of inferior vena cava collapsibility/caval index (ICV CI), end-point septal separation (EPSS) for determining left ventricular ejection fraction (LVEF), cardiac output determination (stroke volume x heart rate), stroke volume variation, & radial artery resistance index) augments standard vital sign assessment (pulse pressure and systolic / diastolic predominance) in clinical decision-making potentially leading to more appropriate pharmacologic and clinical therapies with faster resolution of severe hypertension among pregnant women and women in the postpartum period.

DETAILED DESCRIPTION:
* Minutes count when it comes to treating and preventing serious complications associated with hypertensive emergencies in pregnancy. The rates of maternal morbidity and mortality are on the rise within the United States whereas the rates are falling in the rest of the developed world. Cardiovascular and neurologic injury associated with the severe hypertension witnessed among women with preeclampsia/eclampsia represent two of the leading causes of maternal mortality within the U.S. Optimizing the clinical identification and response to these perinatal complications represents one means of reducing overall maternal mortality.
* Point-of-care use of ultrasound technology to augment clinical diagnosis and management is gaining traction throughout nearly all fields of medicine. Obstetricians utilize this technology frequently to assess the fetus and maternal-fetal interface, and our ability to expand its use to assess a deeper understanding of maternal physiology is underutilized. Exploration into the ability to apply clinically-proven point-of-care sonographic techniques to augment maternal care and reduce maternal mortality is warranted.
* The purpose of this study is to gain a deeper understanding of maternal physiologic changes using easily-obtainable sonographic vascular measurements in the setting of hypertensive emergencies and to assess the utility of these adjunctive maternal sonographic measurements in augmenting clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* For symptomatic women, those presenting to triage, admitted to Labor & Delivery or any of the above units who are at risk for developing a hypertensive emergency will be identified by the OBGYN resident staff or attending physicians as "at risk" for hypertensive emergency as based on current chronic hypertension, gestational hypertension, or preeclampsia). Women presenting with or developing new onset hypertensive emergency can be offered recruitment as well given that the performance of these sonographic measures will not interfere with initiating antihypertensive therapy.

Exclusion Criteria:

* Age < 18 years
* Non-pregnant
* Without the capacity to provide informed written consent
* Non-English speaking without the ability to obtain a hospital interpreter
* Known atrial-ventricular heart block
* History of heart failure
* Moderate-to-Severe bronchial asthma
* Allergy to the medications used as part of regular care treatment of the patient population
* Lack of intravenous IV access
* Concurrent use of antihypertensive medications
* Congenital heart disease in the mother

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Group 1: All pregnant women (under the care of the Maternal-Fetal Medicine physicians or Faculty Medical Center physicians with MFM involvement) experiencing a hypertensive emergency (sustained systolic blood pressure > 160 mmHg or sustained diastolic blood pressure > 110 mmHg {or both} on at least two consecutive occasions 15 minutes apart). All participants must be over the age of 18 and capable of consenting to the study (conscious, with capacity for medical decision making for themselves).
  * Group 2: All asymptomatic pregnant women who are undergoing routine obstetric ultrasound evaluations at any gestational age who elect to undergo cardiovascular sonographic assessment for research purposes at no cost. All participants must be over the age of 18 and capable of consenting to the study (conscious, with capacity for medical decision making for themselves).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | At Enrollment into the Study
  Systolic Blood Pressure at Enrollment into the Study

CONTACTS AND LOCATIONS:
Overall Officials: William Schnettler, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth - Good Samaritan and Bethesda North Hospitals, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No